CLINICAL TRIAL: NCT03416673
Title: Clinical Effectiveness of Coronally Advanced Flap With Papillary Extended Connective Tissue Graft Versus Connective Tissue Graft in Miller Class III Recession: A Randomized Clinical Trial
Brief Title: Effectiveness of the Papillary Extended Connective Tissue Graft in Miller Class III Gingival Recession
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar El-Zanaty, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: peCTG-MC3
Record Dates: First submitted 2018-01-18; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTG+CAF (Active Comparator): The surgical procedure will include a connective tissue graft harvested from the palate and used under a coronally advanced flap
  Interventions: Procedure: CTG+CAF
- peCTG+CAF (Experimental): A papillary extended connective tissue graft reshaped after harvested from the palate will be used under a coronally advanced flap
  Interventions: Procedure: peCTG+CAF

INTERVENTIONS:
Procedure: peCTG+CAF — A connective tissue graft will be reshaped to have extensions mimicking the papillae to augment the inter-dental papillae recessed
  Arms: peCTG+CAF
Procedure: CTG+CAF — A connective tissue graft harvested from the palate will be sutured to the gingival recession site and covered with a coronally advanced flap
  Arms: CTG+CAF

SUMMARY:
34 patients with Miller class III will be included in this study, where 17 participants will be treated with connective tissue graft with coronally advanced flap (control group) and 17 participants will be treated with a papillary extended connective tissue graft with coronally advanced flap (test group) and followed up for 6 months.

DETAILED DESCRIPTION:
Each patient will be inspected to check if the patient fits for the eligibility criteria. If the patient meets the standards, phase I therapy for periodontal plastic procedures will be performed including thorough supragingival scaling and subgingival debridement. Preservation of appropriate plaque control (both mechanical and chemical) by the patient will be executed as well.

Surgical procedures:

It will be done by the principal investigator.

CTG harvesting:

A measurement of the approximate length and width of the graft required will be taken. A CTG will be harvested from the palate using single incision technique as described by Kumar et al. (2013) as follows:

The graft will be harvested from the palate between the distal aspect of the canine and the mid-palatal region of the first molar.

* A template will be placed on the palate to mark the extent of the graft, after local anesthesia is administered.
* A single incision 2 mm apical to the gingival margin will be done. The blade will be placed approximately parallel to the long axis of the palate to provide the first incision.
* The partial thickness flap will be raised as far apically as required, in accordance with the graft size, as measured by the template, using a periosteal elevator. The thickness of the flap will be sufficient to reduce the probability of tearing and sloughing.
* Following this, the blade will be angled perpendicular to the palate through the same incision and continued to the bone. After the incision to the bone, the connective tissue will be elevated from the underlying bone with a periosteal elevator. Then two vertical incisions on the mesial and distal ends of the graft and one horizontal medial incision will be performed (under the partial thickness flap), to release it from the surrounding tissue.
* The graft will be harvested through that single incision and pressure applied to the donor site with gauze soaked in saline after the graft was taken. The donor site will be sutured using a 4-0 silk suture.

For the peCTG, the CTG will be furtherly prepared by creating the papillary extensions using a tissue punch, according to the number of teeth with gingival recession.

Surgical protocol:

The surgical area will be prepared and adequately anesthetized using 4% articaine hydrochloride 1/100 000 epinephrine by giving block and/or infiltration anesthesia. After attaining adequate anesthesia, at a point apical to the papilla tip, vertical incisions will be made lateral to the area of recession extending into alveolar mucosa. The alveolar mucosa between the two vertical incisions will then be undermined by sharp dissection with undermining going into the vestibule while remaining parallel with the surface. Then, a sulcular incision will be used to reflect the coronal portion of the flap by sharp dissection close to the periostium until reaching the split thickness incision

previously made in alveolar mucosa. A gingivoplasty of each papilla adjacent to the recession will then be performed. This excision will not reduce the height of the papilla, but is designed to create a bleeding surface which will serve as a bed for the connective tissue graft (Allen and Miller, 1989).

A triangular flap will be elevated by a sharp dissection with no. 15c scalpel blade to raise a combined full-partial thickness flap to the level of the MGJ.

In the test group (group A), peCTG will be placed over the recession defect leaving the coronal margin of the graft at the level of the CEJ, and the papillary extensions are inserted interdentally covering the de-epithelized papillae, while in the control group (group B), CTG will be also placed over the recession defect leaving the coronal margin of the graft at the level of the CEJ. In both groups, all graft material will be sutured to the periosteum using 6-0 resorbable suture. Finally the flaps will be positioned coronally to the CEJ without tension using 6-0 polyglycolic acid suture material. Hemostasis will be achieved by applying gentle finger pressure for 4 minutes.

Post-surgical protocol:

* Postoperative oral analgesics (Ibuprofen 600 mg t.d.s) will be prescribed to the patients for the first 3 days then whenever desirable. Systemic antibiotic will be prescribed (Amoxicillin 500mg t.d.s) for 5 days to prevent the infection postsurgical.
* Patients will be instructed to rinse with 0.12% Chlorhexidine oral rinse twice daily for 2 weeks.
* Participants will be instructed to avoid excessive muscle tractioning or trauma to the treated areas for the first 3 weeks and will be told not to brush teeth involved in the surgery.
* After 10-14 days the sutures will be removed.
* Three weeks post surgically the patients will be instructed to gently brush the operated area with a soft tooth brush using roll technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older. Periodontally and systemically healthy. Buccal recession defects classified as Miller class III. Presence of identifiable CEJ (Zucchelli et al., 2010). Clinical indication and/or patient demand for recession coverage. O'Leary index less than 20% (O'Leary et al., 1972).

Exclusion Criteria:

* Miller class I, II or IV recession defects. Pregnant females. Smokers as smoking is contraindicated at any plastic periodontal surgery (Khuller, 2009).

Handicapped and mentally retarded patients. Teeth with cervical restorations or abrasion. Taking medication known to affect periodontal healing. Previous periodontal surgery on the involved site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Recession Depth in mm | 6 months
  The vertical amount of root exposed will be measured using a UNC-15 periodontal probe

SECONDARY OUTCOMES:
Recession Width in mm | 6 months
  The width of the exposed root will be measured using a UNC-15 periodontal probe
Probing depth in mm | 6 months
  Measured from the gingival margin to the base of the sulcus will be measured using a UNC-15 periodontal probe
Gingival thickness in mm | 6 months
  the thickness of the gingival tissues will be measured by piercing the gingiva till touching bone with a #15 endodontic reamer under anethesia
Width of keratinized gingiva in mm | 6 months
  from the gingival margin to the mucogingival junction will be measured using a UNC-15 periodontal probe
Root coverage esthetic score (Cairo et al. 2009) | 6 months
  evaluation of the esthetic outcomes of root coverage procedures according to Cairo et al. 2009 Root Coverage Esthetic Score
Patient satisfaction (Kim et al. 2014) | 6 months
  measuring the degree of satisfaction of the patients according to Kim et al. 2014 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Manar T Elzanaty, Master, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cairo F, Cortellini P, Tonetti M, Nieri M, Mervelt J, Cincinelli S, Pini-Prato G. Coronally advanced flap with and without connective tissue graft for the treatment of single maxillary gingival recession with loss of inter-dental attachment. A randomized controlled clinical trial. J Clin Periodontol. 2012 Aug;39(8):760-8. doi: 10.1111/j.1600-051X.2012.01903.x. Epub 2012 May 28. PMID 22639845
- [Background] Chambrone L, Tatakis DN. Periodontal soft tissue root coverage procedures: a systematic review from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S8-51. doi: 10.1902/jop.2015.130674. PMID 25644302
- [Background] Kumar A, Sood V, Masamatti SS, Triveni MG, Mehta DS, Khatri M, Agarwal V. Modified single incision technique to harvest subepithelial connective tissue graft. J Indian Soc Periodontol. 2013 Sep;17(5):676-80. doi: 10.4103/0972-124X.119294. PMID 24174767
- [Background] Cairo F, Rotundo R, Miller PD, Pini Prato GP. Root coverage esthetic score: a system to evaluate the esthetic outcome of the treatment of gingival recession through evaluation of clinical cases. J Periodontol. 2009 Apr;80(4):705-10. doi: 10.1902/jop.2009.080565. PMID 19335093